CLINICAL TRIAL: NCT01692522
Title: Comparison of the Pediatric Intubation on Laryngeal Masks Ambu Aira-i and AirQ for Simulated Blind Intubation in Anesthetized Children
Brief Title: Comparison of the Laryngeal Mask Ambu Aura-i Versus AirQ in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Principal Investigator, Lorenz Theiler, Principal Investigator, Insel Gruppe AG, University Hospital Bern
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: 093/12
Record Dates: First submitted 2012-09-17; First posted 2012-09-25 (Estimated); Last update posted 2014-08-18 (Estimated); Status verified 2014-08

CONDITIONS: Intubation; Difficult
MeSH Terms: interventions — Intubation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ambu Aura-i (Experimental): intubation
  Interventions: Procedure: Intubation
- AirQ (Active Comparator): intubation
  Interventions: Procedure: Intubation

INTERVENTIONS:
Procedure: Intubation — visualized blind intubation

SUMMARY:
The investigators will evaluate the first attempt visualized blind intubation through an Ambu Aura-i versus an AirQ.

DETAILED DESCRIPTION:
After induction of anesthesia, one of the 2 laryngeal masks (Ambu or AirQ) is going to be inserted. Following this, a tracheal tube is mounted on a fiberoptic scope with the tip of the scope behind the tip of the tube. This way, the tracheal tube is not guided by the scope, but the scope visualizes the course of the tracheal tube in the laryngeal mask and the glottic opening as if the tracheal tube was advanced blindly: Visualized blind intubation

ELIGIBILITY:
Inclusion Criteria:

* 0-16 years
* max 50kg
* ASA I-III

Exclusion Criteria:

* risk of aspiration
* known difficult airway
* congenital malformations respiratory tract

Max Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2012-10; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
First attempt visualized blind intubation success rate | how many seconds needed

SECONDARY OUTCOMES:
Overall intubation success rate | how many seconds needed

CONTACTS AND LOCATIONS:
Overall Officials: Robert Greif, MD MME FERC, Study Chair — University Dept Anesthesiology and Pain Therapy, University of Berne, Switzerland
Locations (1):
- Bern University Hospital, Bern, Canton of Bern, Switzerland

REFERENCES:
- [Derived] Kleine-Brueggeney M, Nicolet A, Nabecker S, Seiler S, Stucki F, Greif R, Theiler L. Blind intubation of anaesthetised children with supraglottic airway devices AmbuAura-i and Air-Q cannot be recommended: A randomised controlled trial. Eur J Anaesthesiol. 2015 Sep;32(9):631-9. doi: 10.1097/EJA.0000000000000261. PMID 26061874